CLINICAL TRIAL: NCT05347459
Title: Investigating the Protective Effect of Newer Antidiabetic Drugs on Cognitive Decline in Diabetic Patients
Brief Title: Cognitive Protective Effect of Newer Antidiabetic Drugs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed El-Yazbi, Professor, Alexandria University
Other Study IDs: DIAB-DRUG-COG-FUN-1
Record Dates: First submitted 2022-01-20; First posted 2022-04-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; empagliflozin; Canagliflozin; Sitagliptin Phosphate; saxagliptin; Linagliptin; Vildagliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- New Antidiabetic: Type 2 diabetic patients receiving SGLT2 inhibitors and/or DPP-4 inhibitors with metformin
  Interventions: Drug: Dapagliflozin; Drug: Empagliflozin; Drug: Canagliflozin; Drug: Sitagliptin; Drug: Saxagliptin; Drug: Linagliptin; Drug: Vildagliptin
- Traditional Antidiabetic: Type 2 diabetic patients treated with metformin
- Control: Healthy non-diabetic patients

INTERVENTIONS:
Drug: Dapagliflozin — usual and customary doses for type 2 diabetes management
  Groups: New Antidiabetic
Drug: Empagliflozin — usual and customary doses for type 2 diabetes management
  Groups: New Antidiabetic
Drug: Canagliflozin — usual and customary doses for type 2 diabetes management
  Groups: New Antidiabetic
Drug: Sitagliptin — usual and customary doses for type 2 diabetes management
  Groups: New Antidiabetic
Drug: Saxagliptin — usual and customary doses for type 2 diabetes management
  Groups: New Antidiabetic
Drug: Linagliptin — usual and customary doses for type 2 diabetes management
  Groups: New Antidiabetic
Drug: Vildagliptin — usual and customary doses for type 2 diabetes management
  Groups: New Antidiabetic

SUMMARY:
The proposed study aims to:

1. Explore the cognitive protective effects of SGLT2 inhibitors and DPP-4 inhibitors in patients attending diabetic clinics in Alexandria
2. Examine the possible relationship of such effects with the systemic inflammatory and metabolic status in these patients
3. Undertake a network analysis to elucidate the potential pathways linking the observed protective effects, if any, with the observed changes in inflammatory or metabolic parameters

DETAILED DESCRIPTION:
The investigators propose to profile diabetic patients taking SGLT2 inhibitors and DPP-4 inhibitors using different parameters and compare them to others on more traditional anti-diabetic therapy. Regression and comparative statistics will be used to determine whether the targeted drug classes offer a benefit in terms of cognitive function. If a trend (or correlation) is determined, a bioinformatic approach will be adopted to perform a network analysis including the targets of these drug classes and pathways showing in datasets of the inflammatory or metabolic parameters altered by the drug. This network analysis is intended to provide further mechanistic insight into the pathways involved in the observed drug action.

The patients targeted will be divided into the following groups:

1. Diabetic patients treated with metformin and DPP-4 inhibitors and/or SGLT2 inhibitors
2. Diabetic patients treated with metformin only

This will be in addition to a group of healthy non-diabetic controls to serve as a baseline reference.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetic Patients
* Age (≥50 Years)
* Ability to understand and cooperate with study procedures

Exclusion Criteria:

* Diagnosed dementia
* Use of possible or known cognition impairing drugs in the last three months

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetic patients receiving care in diabetes ambulatory clinics in Alexandria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Prevention of decline in cognitive function associated with type 2 diabetes | 1 Year
  Slowed reduction of the Montreal Cognitive Assessment Battery Score

SECONDARY OUTCOMES:
Better cognitive performance in the intervention group at baseline | 1 Year
  Higher Montreal Cognitive Assessment Battery Score

OTHER OUTCOMES:
Reduced serum inflammatory markers in intervention group | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed F El-Yazbi, PhD, Principal Investigator — Professor of Pharmacology and Therapeutics, Alexandria University; Labiba El-Khordagui, PhD, Principal Investigator — Professor of Pharmaceutics, Alexandria University; Noha A Hamdy, PhD, Principal Investigator — Assistant Professor of Clinical Pharmacy, Alexandria University; Amr El-Feky, MD, Principal Investigator — Assistant Professor of Internal Medicine, Alexandria University; Shams T Osman, BPharm, Principal Investigator — Instructor of Clinical Pharmacy, Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After publication a link will be provided for a data repository folder
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be come available after publication and remain available indefinitely
Access Criteria: Anyone who wishes to access the data